CLINICAL TRIAL: NCT03175367
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Varying Doses and Dose Regimens of Evinacumab in Patients With Persistent Hypercholesterolemia Despite Maximally Tolerated Lipid Modifying Therapy
Brief Title: Study of Evinacumab (REGN1500) in Participants With Persistent Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R1500-CL-1643; 2017-001508-31 (EudraCT Number)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group A: dosing regimen 1 (Experimental): SC Evinacumab QW for 16 weeks
  Interventions: Drug: Evinacumab; Other: Background Lipid Modifying Therapy (LMT)
- Group A: dosing regimen 2 (Experimental): SC Evinacumab Q2W for 16 weeks (alternating with matching placebo on opposite weeks)
  Interventions: Drug: Evinacumab; Other: Background Lipid Modifying Therapy (LMT)
- Group A: dosing regimen 3 (Experimental): SC Evinacumab QW for 16 weeks
  Interventions: Drug: Evinacumab; Other: Background Lipid Modifying Therapy (LMT)
- Group A: matching placebo (Experimental): Placebo SC QW for 16 weeks
  Interventions: Drug: Matching placebo; Other: Background Lipid Modifying Therapy (LMT)
- Group B: dosing regimen 1 (Experimental): Intravenous (IV) Evinacumab Q4W for 24 weeks
  Interventions: Drug: Evinacumab; Other: Background Lipid Modifying Therapy (LMT)
- Group B: dosing regimen 2 (Experimental): IV Evinacumab Q4W for 24 weeks
  Interventions: Drug: Evinacumab; Other: Background Lipid Modifying Therapy (LMT)
- Group B: matching placebo (Experimental): Placebo IV Q4W for 24 weeks
  Interventions: Drug: Matching placebo; Other: Background Lipid Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Evinacumab — SC or IV administration
  Other Names: REGN1500
  Arms: Group A: dosing regimen 1; Group A: dosing regimen 2; Group A: dosing regimen 3; Group B: dosing regimen 1; Group B: dosing regimen 2
Drug: Matching placebo — SC or IV administration
  Arms: Group A: matching placebo; Group B: matching placebo
Other: Background Lipid Modifying Therapy (LMT) — All participants should be on a stable, maximally tolerated statin throughout the duration of the study. The dose of statin and of PCSK9 inhibitor, such as alirocumab or evolocumab, as well as other LMT (if applicable), should remain stable throughout the study duration, from screening through the end of study (EOS) visit.

SUMMARY:
The primary objective of the study is to evaluate the reduction of LDL-C by evinacumab in comparison to placebo after 16 weeks in patients with primary hypercholesterolemia (HeFH, or non-HeFH with a history of clinical ASCVD) with persistent hypercholesterolemia despite receiving maximally-tolerated LMT. Persistent hypercholesterolemia is defined as LDL-C ≥70 mg/dL (1.81 mmol/L) for those patients with clinical ASCVD and LDL-C ≥100 mg/dL (2.59 mmol/L) for those patients without clinical ASCVD.

ELIGIBILITY:
The inclusion/ exclusion criteria below, include, but are not limited to, the following:

Key Inclusion Criteria:

1. Men and women, ages 18 through 80 at the screening visit
2. Diagnosis of primary hypercholesterolemia, either HeFH or non-HeFH with clinical ASCVD
3. A history of clinical ASCVD, for those patients who are non-HeFH.
4. Receiving a stable maximally tolerated statin (± ezetimibe) for at least 4 weeks at screening
5. For those patients with HeFH who are not receiving a statin at screening, documentation of inability to tolerate at least 2 statins.
6. Receiving alirocumab 150 mg SC Q2W, OR evolocumab 140 mg SC Q2W or 420 mg SC Q4W for at least 8 weeks prior to the screening visit
7. For those patients with a history of clinical ASCVD, serum LDL-C ≥ 70 mg/dL at screening (1 repeat lab is allowed)
8. For those patients without a history of clinical ASCVD, serum LDL-C ≥ 100 mg/dL at screening (1 repeat lab is allowed)
9. Provide signed informed consent

Key Exclusion Criteria:

1. Known history of homozygous FH (clinically, or by previous genotyping)
2. Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins
3. Newly diagnosed diabetes (within 3 months prior to screening)
4. Use of thyroid medications (except for replacement therapy which has been stable for at least 12 weeks before screening)
5. Laboratory findings during screening period (not including randomization labs):

   1. Triglycerides > 400 mg/dL (> 4.52 mmol/L) for patients without a known history of diabetes mellitus; OR Triglycerides > 300 mg/dL (> 3.39 mmol/L) for patients with a known history of diabetes mellitus
   2. Positive test for Hepatitis B surface antigen and/or Hepatitis C antibody (associated with a positive HCV ribonucleic acid [RNA] polymerase chain reaction)
   3. Positive serum beta-human chorionic gonadotropin or urine pregnancy test in women of childbearing potential
   4. Estimated glomerular filtration rate < 30 mL/min/1.73 m^2
   5. TSH > 1.5 x ULN
   6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x ULN
6. Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at screening visit or time of randomization
7. History of heart failure (New York Heart Association [NYHA] Class III-IV) within 12 months before screening
8. History of MI, unstable angina leading to hospitalization, CABG surgery, PCI, uncontrolled cardiac arrhythmia, carotid surgery or stenting, stroke, TIA, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease within 3 months prior screening
9. History of cancer within the past 5 years (except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer)
10. Having received LDL apheresis within 2 months before screening
11. Pregnant or breast-feeding women
12. Women of childbearing potential who are unwilling to practice a highly effective birth control method
13. Men who are sexually active with women of childbearing potential (WOCBP) and are unwilling to consistently use condoms during the study drug treatment period regardless of vasectomy status.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (95):
- United States (23):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Office of Dr. John D Homan MD, Newport Beach, California
  - Preventive Cardiology Inc, Boca Raton, Florida
  - Care Research Center Inc, Doral, Florida
  - Florida Lipid Institute, Winter Park, Florida
  - St. Vincent Medical Group, Inc, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - EMMC Northeast Cardiology Assocites, Bangor, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Heart Health Cardiology, Grand Rapids, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mt Sinai Ichan Medical Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rowan Diagnostic Clinic, Salisbury, North Carolina
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - The University Of Texas Health Science Center Houston, Houston, Texas
  - San Antonio Premiere Internal Medicine, San Antonio, Texas
  - Clear Clinical Research, LLC, Schertz, Texas
  - PharmaTex Research, Tyler, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland
- Austria (2):
  - University Hospital Innsbruck - Tyrolean Hospital, Innsbruck, Tyrol
  - Medizinische Universitaetsklinik Graz, Graz
- Canada (4):
  - Robarts Research Institute, London, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Centre Etudes Cliniques Econogene-21, Chicoutimi, Quebec
  - Clinique des maladies lipidiques de Quebec, Québec, Quebec
- Czechia (4):
  - CCR Prague, S.R.O, Prague, Prague 3
  - Univerzita Karlova v Praze 1 Lekarska Fakulta, Karlov, Praha 2
  - University Hospital, Charles University, Hradec Králové
  - Ikem Institut Klinicke A Experimentalni Mediciny, Prague
- Denmark (2):
  - Sydvestjysk Sygehus, Esbjerg
  - Regionshospitalet Herning, Herning
- France (2):
  - Hopital G Et R Laennec, Nantes, Cedex
  - Houpital Du Bocage, Dijon
- Israel (4):
  - Edith Wolfson Medical Center, Holon
  - Galilee Medical Center, Nahariya
  - Sheba Mc, Ramat Gan
  - Sourasky Medical Center, Cardiovascular Research Center, Tel Aviv
- Italy (4):
  - Azienda Ospedaliero Universitaria Federico II di Napoli, Napoli
  - Fondazione Toscana Gabriele Monasterio Per La Ricerca Medica E Di Sanita Pubblica, Pisa
  - Ausl Della Romagna-Ospedale Degli Infermi, Rimini
  - Dipartimento di Medicina Traslazionale e di Precisione dell'Università degli Studi di, Rome
- Japan (4):
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa-shi
  - Minamino Cardiovascular Hospital, Hachiōji
  - Saitama Medical University Hospital, Iruma-gun
- Jordan (4):
  - Istishari Hospital, Amman
  - King Abdullah University Hospital-1, Irbid
  - King Abdullah University Hospital-2, Irbid
  - King Abdullah University Hospital, Irbid
- Netherlands (4):
  - VOC Hoorn, Hoorn, Hoorn Noord-Hollan
  - Admiraal de Ruyter Ziekenhuis, Goes, Zeeland
  - Academic Medical Center, Amsterdam
  - Universitair Medisch Centrum Utrech - Locatie AZU, Utrecht
- New Zealand (3):
  - Lipid and Diabetes Research Group, Christchurch, Canterbury
  - Papamoa Pines Medical Centre, Papamoa
  - Clinical Horizons NZ Ltd, Tauranga
- M3 Helse AS, Oslo, Norway
- Poland (4):
  - Halina Serafin NZOZ Centrum Medyczne SERAFIN-MED, Żarów, Lower Silesian Voivodeship
  - Nzoz Przychodnia Specjalistyczna, Ruda Slaska, Podlaskie Voivodeship
  - Wojewodzki Szpital Specjalistyczny, Bytom
  - Slaskie Centrum Chorob Serca, III Katedra i Oddzial Kliniczny Kardiologii SUM- Oddzial Chorob Serca i Naczyn, Zabrze
- Russia (11):
  - Federal State Budgetary Institution Research Institute for Complex Issues of Cardiovacsular Disease, Kemerovo
  - National Research Center For Preventative Medicine of Federal Agency of High Technology Medical Aid, Moscow
  - Federal State Budget Institution Out-patient Clinic 3, Moscow
  - NII of Therapy and Preventive Medicine, Novosibirsk
  - Municipal Medical and Prophylactic Institution - City Hospital for Emergency Care No.2, Rostov-on-Don
  - Limmited Liability Company International Medical Centre SOGAZ, Saint Petersburg
  - Federal State Institution of Healthcare Clinical Hospital #122 N.A.L.G Sokolov, Saint Petersburg
  - LLC- Institute of Medical Research, Saint Petersburg
  - Federal State Budgetary Institution Clinical-Diagnostic Center with Polyclinic, Saint Petersburg
  - Samara Regional Clinical Cardiologic Dispensary, Samara
  - Cardiology Research Institute, Tomsk
- South Africa (5):
  - The Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Jongaie Research, Pretoria, West Gauteng
  - Dr JM Engelbrecht Trial Site, Cape Town, Western Cape
  - University of Cape Town, Cape Town
  - TREAD Research CC, Parow
- Spain (6):
  - Hospital Universitario A Coruna, A Coruña, A Coruna
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves (HUVN), Granada
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (4):
  - Karolinska University Hospital, Malmo
  - Akardo MedSite, Stockholm
  - Karolinska Institutet, Stockholm
  - Akademiska sjukhuset, Uppsala
- United Kingdom (2):
  - Royal Free Hospital-Royal Free London NHS Foundation Trust, London
  - Royal Victoria Infirmary - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Derived] Rosenson RS, Burgess LJ, Ebenbichler CF, Baum SJ, Stroes ESG, Ali S, Khilla N, McGinniss J, Gaudet D, Pordy R. Longer-Term Efficacy and Safety of Evinacumab in Patients With Refractory Hypercholesterolemia. JAMA Cardiol. 2023 Nov 1;8(11):1070-1076. doi: 10.1001/jamacardio.2023.2921. PMID 37703006
- [Derived] Rosenson RS, Burgess LJ, Ebenbichler CF, Baum SJ, Stroes ESG, Ali S, Khilla N, Hamlin R, Pordy R, Dong Y, Son V, Gaudet D. Evinacumab in Patients with Refractory Hypercholesterolemia. N Engl J Med. 2020 Dec 10;383(24):2307-2319. doi: 10.1056/NEJMoa2031049. Epub 2020 Nov 15. PMID 33196153

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 327 participants were screened and 272 participants randomized. Six participants were randomized but never treated.
Groups:
- Group A: Placebo SC QW (DBTP): Placebo subcutaneous (SC) treatment every week (QW) for 16 weeks during the double-blind treatment period (DBTP) followed by a 23-week follow-up period
- Group A: Evinacumab 300 mg SC Q2W (DBTP): Evinacumab 300 mg SC treatment every other week (Q2W) (alternating with placebo on opposite weeks) for 16 weeks during the DBTP followed by a 23-week follow-up period
- Group A: Evinacumab 300 mg SC QW (DBTP): Evinacumab 300 mg SC treatment QW for 16 weeks during the DBTP followed by a 23-week follow-up period
- Group A: Evinacumab 450 mg SC QW (DBTP): Evinacumab 450 mg SC treatment QW for 16 weeks during the DBTP followed by a 23-week follow-up period
- Group B: Placebo IV Q4W (DBTP to OLTP): Placebo intravenous (IV) treatment every 4 weeks (Q4W) during the DBTP followed by evinacumab 15 mg/kg IV Q4W for a 48-week open-label treatment period (OLTP) regardless of treatment assignment in the DBTP
- Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP): Evinacumab 5 mg/kg IV treatment Q4W during the 24-week DBTP followed by evinacumab 15 mg/kg IV Q4W for a 48-week OLTP regardless of treatment assignment in the DBTP
- Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP): Evinacumab 15 mg/kg IV treatment Q4W during the DBTP followed by evinacumab 15 mg/kg IV Q4W for a 48-week OLTP regardless of treatment assignment in the DBTP
Period: Double-blind Treatment Period (DBTP)
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Started | 39 | 39 | 42 | 40 | 33 | 35 | 38
Completed | 30 | 31 | 30 | 30 | 31 | 32 | 34
Not Completed | 9 | 8 | 12 | 10 | 2 | 3 | 4
Not completed — Protocol Violation | 0 | 0 | 1 | 2 | 0 | 0 | 2
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 2 | 0 | 1 | 0
Not completed — Physician Decision | 6 | 5 | 8 | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Open-Label Treatment Period (OLTP)
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Started (Treated in OLTP) | 0 | 0 | 0 | 0 | 31 | 32 | 33 (One participant completed DBTP, but did not continue to OLTP)
Completed (Completed Study) | 0 | 0 | 0 | 0 | 31 | 30 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Noncompliance with protocol | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP) | Total
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38 | 266
Age, Customized [Number; unit: Participants]
  Adults (18-64 years) | 34 | 29 | 34 | 30 | 26 | 28 | 33 | 214
  From 65-84 years | 5 | 10 | 8 | 10 | 7 | 7 | 5 | 52
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 23 | 29 | 18 | 22 | 19 | 159
  Male | 12 | 18 | 19 | 11 | 15 | 13 | 19 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 2 | 3 | 7 | 2 | 23
  Not Hispanic or Latino | 36 | 31 | 38 | 38 | 30 | 28 | 36 | 237
  Unknown or Not Reported | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 6
  White | 34 | 34 | 39 | 38 | 27 | 32 | 35 | 239
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 3 | 1 | 3 | 2 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol (LDL-C) at Week 16 (Intent-to-Treat [ITT] Estimand)
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percent Change | 8.8 (6.4) [lower limit 6.4] | -29.7 (6.4) [lower limit 6.4] | -44.0 (6.3) [lower limit 6.3] | -47.2 (6.2) [lower limit 6.2] | 0.6 (6.6) [lower limit 6.6] | -23.5 (6.6) [lower limit 6.6] | -49.9 (6.1) [lower limit 6.1]
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -38.5, 95% CI 2-sided [-56.5 to -20.6], Standard Error of Mean 9.1
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -52.9, 95% CI 2-sided [-70.7 to -35.1], Standard Error of Mean 9.0
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -56.0, 95% CI 2-sided [-73.7 to -38.3], Standard Error of Mean 9.0
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0109, Mixed Models Analysis — P-Value is not adjusted for multiplicity; Least Squares Mean Difference = -24.2, 95% CI 2-sided [-42.6 to -5.7], Standard Error of Mean 9.3
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -50.5, 95% CI 2-sided [-68.4 to -32.6], Standard Error of Mean 9.0

2. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 16 (ITT Estimand)
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percent Change | 6.7 (5.1) [lower limit 5.1] | -19.9 (5.1) [lower limit 5.1] | -35.2 (5.1) [lower limit 5.1] | -38.8 (4.9) [lower limit 4.9] | -3.8 (4.7) [lower limit 4.7] | -20.4 (4.6) [lower limit 4.6] | -43.2 (4.3) [lower limit 4.3]
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p = 0.0003, Mixed Models Analysis; Least Squares Mean Difference = -26.6, 95% CI 2-sided [-40.9 to -12.4], Standard Error of Mean 7.2
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -42.0, 95% CI 2-sided [-56.1 to -27.9], Standard Error of Mean 7.1
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -45.5, 95% CI 2-sided [-59.5 to -31.5], Standard Error of Mean 7.1
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0132, Mixed Models Analysis; Least Squares Mean Difference = -16.6, 95% CI 2-sided [-29.7 to -3.5], Standard Error of Mean 6.6
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -39.4, 95% CI 2-sided [-52.0 to -26.8], Standard Error of Mean 6.4

3. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 (ITT Estimand)
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 33 | 35 | 38
Percent Change | 5.9 (6.0) [lower limit 6.0] | -15.9 (5.9) [lower limit 5.9] | -34.5 (5.6) [lower limit 5.6]
Statistical Analysis 1: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0111, Mixed Models Analysis; Least Squares Mean Difference = -21.8, 95% CI 2-sided [-38.4 to -5.1], Standard Error of Mean 8.4
Statistical Analysis 2: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -40.4, 95% CI 2-sided [-56.7 to -24.0], Standard Error of Mean 8.2

4. Secondary Outcome: Percent Change From Baseline in Non High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 16 (ITT Estimand)
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percent Change | 8.0 (5.4) [lower limit 5.4] | -31.3 (5.4) [lower limit 5.4] | -45.8 (5.3) [lower limit 5.3] | -50.6 (5.2) [lower limit 5.2] | -1.1 (5.8) [lower limit 5.8] | -24.8 (5.7) [lower limit 5.7] | -52.0 (5.3) [lower limit 5.3]
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -39.3, 95% CI 2-sided [-54.4 to -24.3], Standard Error of Mean 7.6
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -53.8, 95% CI 2-sided [-68.8 to -38.9], Standard Error of Mean 7.6
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -58.5, 95% CI 2-sided [-73.4 to -43.7], Standard Error of Mean 7.5
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0042, Mixed Models Analysis; Least Squares Mean Difference = -23.7, 95% CI 2-sided [-39.7 to -7.7], Standard Error of Mean 8.1
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -50.9, 95% CI 2-sided [-66.4 to -35.4], Standard Error of Mean 7.8

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 (ITT Estimand)
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 33 | 35 | 38
Percent Change | 10.4 (7.0) [lower limit 7.0] | -20.2 (6.7) [lower limit 6.7] | -44.3 (6.4) [lower limit 6.4]
Statistical Analysis 1: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0021, Mixed Models Analysis; Least Squares Mean Difference = -30.6, 95% CI 2-sided [-49.8 to -11.4], Standard Error of Mean 9.7
Statistical Analysis 2: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -54.6, 95% CI 2-sided [-73.4 to -35.8], Standard Error of Mean 9.5

6. Secondary Outcome: Percentage of Participants With >= 30% Reduction in Calculated LDL-C at Week 16 (ITT Estimand)
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percentage of Participants | 11.3 | 68.1 | 73.9 | 71.4 | 15.5 | 57.9 | 86.8
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio, log = 19.4, 95% CI 2-sided [5.1 to 72.8]
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio, log = 23.9, 95% CI 2-sided [6.4 to 89.2]
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio, log = 22.1, 95% CI 2-sided [6.0 to 80.5]
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio, log = 8.5, 95% CI 2-sided [2.5 to 29.2]
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio, log = 42.3, 95% CI 2-sided [10.4 to 172.3]

7. Secondary Outcome: Percentage of Participants With >= 50% Reduction in Calculated LDL-C at Week 16 (ITT Estimand)
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percentage of Participants | 5.2 | 28.6 | 53.7 | 60.6 | 12.3 | 24.6 | 63.2
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p = 0.0100, Regression, Logistic; Odds Ratio (OR) = 9.6, 95% CI 2-sided [1.7 to 53.5]
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 24.8, 95% CI 2-sided [4.7 to 129.9]
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 36.1, 95% CI 2-sided [6.7 to 194.7]
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.3185, Regression, Logistic; Odds Ratio (OR) = 2.0, 95% CI 2-sided [0.5 to 8.2]
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 14.5, 95% CI 2-sided [3.9 to 54.2]

8. Secondary Outcome: Percentage of Participants With Calculated LDL-C < 50 mg/dL (1.30 mmol/L) at Week 16 (ITT Estimand)
Description: Percentage of Participants with Calculated LDL-C < 50 milligrams/deciliter (mg/dL) [1.30 Millimoles per liter (mmol/L)] at Week 16 (ITT Estimand)
Time Frame: Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percentage of Participants | 5.1 | 22.8 | 29.7 | 40.8 | 9.3 | 13.2 | 39.5
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p = 0.0718, Regression, Logistic; Odds Ratio (OR) = 4.8, 95% CI 2-sided [0.9 to 26.5]
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p = 0.0048, Regression, Logistic; Odds Ratio (OR) = 11.4, 95% CI 2-sided [2.1 to 62.1]
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p = 0.0015, Regression, Logistic; Odds Ratio (OR) = 14.7, 95% CI 2-sided [2.8 to 76.8]
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.5270, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.3 to 8.4]
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0047, Regression, Logistic; Odds Ratio (OR) = 7.7, 95% CI 2-sided [1.9 to 31.7]

9. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 (ITT Estimand)
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 33 | 35 | 38
Percent Change | 14.8 (8.3) [lower limit 8.3] | -17.7 (8.0) [lower limit 8.0] | -39.7 (7.7) [lower limit 7.7]
Statistical Analysis 1: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0059, Mixed Models Analysis; Least Squares Mean Difference = -32.5, 95% CI 2-sided [-55.5 to -9.6], Standard Error of Mean 11.5
Statistical Analysis 2: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -54.5, 95% CI 2-sided [-77.0 to -32.0], Standard Error of Mean 11.3

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 16 (ITT Estimand)
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percent Change | 6.1 (4.0) [lower limit 4.0] | -31.0 (4.0) [lower limit 4.0] | -40.3 (4.0) [lower limit 4.0] | -45.4 (3.9) [lower limit 3.9] | -0.4 (4.5) [lower limit 4.5] | -22.6 (4.4) [lower limit 4.4] | -46.8 (4.1) [lower limit 4.1]
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -37.1, 95% CI 2-sided [-48.4 to -25.8], Standard Error of Mean 5.7
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -46.4, 95% CI 2-sided [-57.5 to -35.2], Standard Error of Mean 5.6
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -51.5, 95% CI 2-sided [-62.5 to -40.4], Standard Error of Mean 5.6
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0006, Mixed Models Analysis; Least Squares Mean Difference = -22.2, 95% CI 2-sided [-34.6 to -9.8], Standard Error of Mean 6.2
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -46.4, 95% CI 2-sided [-58.4 to -34.4], Standard Error of Mean 6.1

11. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 24 (ITT Estimand)
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 33 | 35 | 38
Percent Change | 8.5 (5.1) [lower limit 5.1] | -19.9 (4.9) [lower limit 4.9] | -40.8 (4.7) [lower limit 4.7]
Statistical Analysis 1: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -28.4, 95% CI 2-sided [-42.6 to -14.3], Standard Error of Mean 7.1
Statistical Analysis 2: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -49.3, 95% CI 2-sided [-63.2 to -35.4], Standard Error of Mean 7.0

12. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 16 (ITT Estimand)
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percent Change | 8.1 (4.5) [lower limit 4.5] | -38.0 (4.2) [lower limit 4.2] | -47.7 (4.0) [lower limit 4.0] | -53.4 (3.9) [lower limit 3.9] | -6.9 (4.7) [lower limit 4.7] | -32.1 (4.5) [lower limit 4.5] | -52.8 (4.1) [lower limit 4.1]
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p < .0001, Regression, Linear; Adjusted Mean Difference = -46.1, 95% CI 2-sided [-57.8 to -34.3], Standard Error of Mean 6.0
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p < .0001, Regression, Linear; Adjusted Mean Difference = -55.8, 95% CI 2-sided [-67.3 to -44.3], Standard Error of Mean 5.9
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p < .0001, Regression, Linear; Adjusted Mean Difference = -61.5, 95% CI 2-sided [-72.9 to -50.0], Standard Error of Mean 5.8
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0001, Regression, Linear; Adjusted Mean Difference = -25.2, 95% CI 2-sided [-38.0 to -12.4], Standard Error of Mean 6.5
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < .0001, Regression, Linear; Adjusted Mean Difference = -45.9, 95% CI 2-sided [-58.4 to -33.5], Standard Error of Mean 6.3

13. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 (ITT Estimand)
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 33 | 35 | 38
Percent Change | -6.1 (5.4) [lower limit 5.4] | -23.2 (5.1) [lower limit 5.1] | -51.3 (4.8) [lower limit 4.8]
Statistical Analysis 1: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0228, Regression, Linear; Adjusted Mean Difference = -17.1, 95% CI 2-sided [-31.8 to -2.4], Standard Error of Mean 7.5
Statistical Analysis 2: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p < .0001, Regression, Linear; Adjusted Mean Difference = -45.3, 95% CI 2-sided [-59.6 to -31.0], Standard Error of Mean 7.3

14. Secondary Outcome: Percent Change From Baseline in Lipoprotein a [Lp(a)] at Week 16 (ITT Estimand)
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 39 | 39 | 42 | 40 | 33 | 35 | 38
Percent Change | 0.3 (3.9) [lower limit 3.9] | -10.3 (4.1) [lower limit 4.1] | -11.6 (4.0) [lower limit 4.0] | -8.9 (4.0) [lower limit 4.0] | 0.8 (3.7) [lower limit 3.7] | -15.7 (3.7) [lower limit 3.7] | -15.7 (3.3) [lower limit 3.3]
Statistical Analysis 1: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC Q2W (DBTP); Test type: Superiority; p = 0.0635, Regression, Linear; Adjusted Mean Difference = -10.6, 95% CI 2-sided [-21.8 to 0.6], Standard Error of Mean 5.7
Statistical Analysis 2: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 300 mg SC QW (DBTP); Test type: Superiority; p = 0.0314, Regression, Linear; Adjusted Mean Difference = -11.9, 95% CI 2-sided [-22.8 to -1.1], Standard Error of Mean 5.5
Statistical Analysis 3: Comparison: Group A: Placebo SC QW (DBTP) vs Group A: Evinacumab 450 mg SC QW (DBTP); Test type: Superiority; p = 0.0923, Regression, Linear; Adjusted Mean Difference = -9.2, 95% CI 2-sided [-19.9 to 1.5], Standard Error of Mean 5.5
Statistical Analysis 4: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0017, Regression, Linear; Adjusted Mean Difference = -16.5, 95% CI 2-sided [-26.8 to -6.2], Standard Error of Mean 5.3
Statistical Analysis 5: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0009, Regression, Linear; Adjusted Mean Difference = -16.5, 95% CI 2-sided [-26.2 to -6.8], Standard Error of Mean 4.9

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) [Lp(a)] at Week 24 (ITT Estimand)
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Group B: Placebo IV Q4W (DBTP to OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP)
Number analyzed (Participants) | 33 | 35 | 38
Percent Change | -1.4 (4.1) [lower limit 4.1] | -17.5 (4.0) [lower limit 4.0] | -16.0 (3.7) [lower limit 3.7]
Statistical Analysis 1: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 5 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0054, Regression, Linear; Adjusted Mean Difference = -16.1, 95% CI 2-sided [-27.4 to -4.7], Standard Error of Mean 5.8
Statistical Analysis 2: Comparison: Group B: Placebo IV Q4W (DBTP to OLTP) vs Group B: Evinacumab 15 mg/kg IV Q4W (DBTP to OLTP); Test type: Superiority; p = 0.0085, Regression, Linear; Adjusted Mean Difference = -14.6, 95% CI 2-sided [-25.4 to -3.7], Standard Error of Mean 5.5

ADVERSE EVENTS:
Time Frame: Group A from day of first treatment up to 39 weeks, Group B from day of first treatment up to 92 weeks
Description: 1 participant randomized to the "Group B: Evinacumab 15 mg/kg IV Q4W (DBTP)" arm inadvertently received evinacumab 5 mg/kg IV at all double-blind administration visits. Per the study statistical analysis plan (SAP), this participant's safety data was analyzed as treated in the "Group B: Evinacumab 5 mg/kg IV Q4W (DBTP)" arm.
Groups:
- Group B: Placebo IV Q4W (DBTP); Group B: Placebo IV Q4W (OLTP): Placebo intravenous (IV) treatment every 4 weeks (Q4W) during the DBTP followed by evinacumab 15 mg/kg IV Q4W for a 48-week open-label treatment period (OLTP) regardless of treatment assignment in the DBTP
- Group B: Evinacumab 5 mg/kg IV Q4W (DBTP); Group B: Evinacumab 5 mg/kg IV Q4W (OLTP): Evinacumab 5 mg/kg IV treatment Q4W during the 24-week DBTP followed by evinacumab 15 mg/kg IV Q4W for a 48-week OLTP regardless of treatment assignment in the DBTP
- Group B: Evinacumab 15 mg/kg IV Q4W (DBTP); Group B: Evinacumab 15 mg/kg IV Q4W (OLTP): Evinacumab 15 mg/kg IV treatment Q4W during the DBTP followed by evinacumab 15 mg/kg IV Q4W for a 48-week OLTP regardless of treatment assignment in the DBTP
Arm/Group | Group A: Placebo SC QW (DBTP) | Group A: Evinacumab 300 mg SC Q2W (DBTP) | Group A: Evinacumab 300 mg SC QW (DBTP) | Group A: Evinacumab 450 mg SC QW (DBTP) | Group B: Placebo IV Q4W (DBTP) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP) | Group B: Placebo IV Q4W (OLTP) | Group B: Evinacumab 5 mg/kg IV Q4W (OLTP) | Group B: Evinacumab 15 mg/kg IV Q4W (OLTP)
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/39 | 1/42 | 0/40 | 0/33 | 0/36 | 0/37 | 0/31 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/39 | 2/39 | 4/42 | 4/40 | 1/33 | 2/36 | 6/37 | 4/31 | 3/32 | 2/33
Other Adverse Events (participants affected / at risk) | 20/39 | 27/39 | 26/42 | 22/40 | 18/33 | 23/36 | 24/37 | 19/31 | 22/32 | 24/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Placebo SC QW (DBTP) (N=39) | Group A: Evinacumab 300 mg SC Q2W (DBTP) (N=39) | Group A: Evinacumab 300 mg SC QW (DBTP) (N=42) | Group A: Evinacumab 450 mg SC QW (DBTP) (N=40) | Group B: Placebo IV Q4W (DBTP) (N=33) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP) (N=36) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP) (N=37) | Group B: Placebo IV Q4W (OLTP) (N=31) | Group B: Evinacumab 5 mg/kg IV Q4W (OLTP) (N=32) | Group B: Evinacumab 15 mg/kg IV Q4W (OLTP) (N=33)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Placebo SC QW (DBTP) (N=39) | Group A: Evinacumab 300 mg SC Q2W (DBTP) (N=39) | Group A: Evinacumab 300 mg SC QW (DBTP) (N=42) | Group A: Evinacumab 450 mg SC QW (DBTP) (N=40) | Group B: Placebo IV Q4W (DBTP) (N=33) | Group B: Evinacumab 5 mg/kg IV Q4W (DBTP) (N=36) | Group B: Evinacumab 15 mg/kg IV Q4W (DBTP) (N=37) | Group B: Placebo IV Q4W (OLTP) (N=31) | Group B: Evinacumab 5 mg/kg IV Q4W (OLTP) (N=32) | Group B: Evinacumab 15 mg/kg IV Q4W (OLTP) (N=33)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 1 (3) | 2 (2) | 4 (5) | 5 (5) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 4 (5) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 2 (4) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (4) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 2 (2) | 3 (5) | 4 (4) | 6 (10) | 2 (3) | 5 (6) | 4 (4) | 2 (2) | 4 (6)
Dizziness (Nervous system disorders) | 5 (6) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 1 (2) | 2 (3) | 3 (17) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 4 (21) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (8) | 3 (3) | 3 (3) | 1 (2) | 1 (1) | 3 (4) | 4 (5)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2) | 4 (15) | 2 (2) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (11) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (4) | 2 (2) | 1 (4) | 4 (26) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 1 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 4 (5) | 4 (5) | 4 (6) | 2 (2) | 3 (4) | 6 (6) | 5 (7) | 4 (4) | 3 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (7) | 5 (6) | 5 (6) | 4 (6) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 6 (8) | 3 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT03175367/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03175367/SAP_001.pdf